CLINICAL TRIAL: NCT00681044
Title: High-Dose Melphalan and Autologous Stem Cell Transplantation (HDM/SCT) in Light-Chain Deposition Disease (LCDD) and Immunoglobulin Deposition Disease (IGDD)
Brief Title: HD Melphalan and SCT in Patients With IGDD or LCDD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Vaishali Sanchorawala, Principal Investigator, Boston Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000595782; BHO-H-25876 (Other); BUMC-H-25876 (Other: Boston University Medical Center IRB)
Record Dates: First submitted 2008-05-18; First posted 2008-05-20 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-03

CONDITIONS: Multiple Myeloma
Keywords: monoclonal immunoglobulin deposition disease; light chain deposition disease
MeSH Terms: conditions — Multiple Myeloma; Immunoglobulin Light-chain Amyloidosis | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCT with melphalan conditioning (Experimental): Mobilization with Filgrastim Stem Cell Transplant Melphalan Conditioning Stem Cell infusion
  Interventions: Biological: filgrastim; Drug: melphalan; Procedure: Stem Cell Infusion

INTERVENTIONS:
Biological: filgrastim — 16 mcg/kg daily beginning 3 days prior to SCC through day before final SCC
  Other Names: G-CSF, neulasta
Drug: melphalan — 70-100 mg/m2/day will be administered intravenously on Days -3 and -2
  Other Names: alkeran
Procedure: Stem Cell Infusion — infusion of previously collected stem cells on Day 0

SUMMARY:
RATIONALE: Giving chemotherapy before a stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as G-CSF, and certain chemotherapy drugs, helps stem cells move from the bone marrow to the blood so they can be collected and stored. Chemotherapy is then given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

PURPOSE: This phase II trial is studying the side effects of high-dose melphalan given together with stem cell transplant and to see how well it works in treating patients with immunoglobulin deposition disease or light-chain deposition disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* To assess the tolerability of high-dose melphalan and autologous stem cell transplantation in patients with immunoglobulin deposition disease or light-chain deposition disease.
* To determine the hematologic response rate in patients treated with this regimen.
* To determine the predictability of early free light-chain response for heme response in patients treated with this regimen.
* To determine organ or clinical response in patients treated with this regimen.
* To determine overall survival of these patients.

OUTLINE:

* Stem cell mobilization: Patients undergo blood stem cell mobilization comprising filgrastim (G-CSF) subcutaneously once daily for 3 days (i.e., through the day before the last stem cell collection).
* Stem cell collection: Patients undergo collection of G-CSF-mobilized blood stem cells until the target number of stem cells (at least 2 x 10^6 cluster of differentiation-34-positive cells) is reached.
* Conditioning regimen: Patients receive high-dose melphalan IV on days -3 to -2.
* Autologous stem cell transplantation: Patients undergo blood stem cell infusion on day 0.

After completion of study therapy, patients are followed at 3, 6, and 12 months and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

DISEASE CHARACTERISTICS:

* Histologically confirmed light-chain deposition disease based on the following criteria:

  * Deposition of granular material containing free light-chain (FLC) immunoglobulins that did not bind Congo red
  * Evidence of a plasma cell dyscrasia, as defined by any of the following:

    * Monoclonal gammopathy in the serum or urine by immunofixation electrophoresis
    * Clonal plasmacytosis on bone marrow biopsy by immuno-histochemical
    * Elevated serum levels of FLC
* Patients may enroll after stem cell collection (SCC) if all prestudy requirements are completed prior to starting SCC (i.e., ≥ 2.5 x 10^6 cells available for transplantation)

PRIOR CONCURRENT THERAPY:

* Prior chemotherapy with alkylating agent allowed provided there is no evidence of myelodysplastic syndromes
* Prior total dose of melphalan < 300 mg
* More than 4 weeks since prior cytotoxic therapy and recovered

PATIENT CHARACTERISTICS:

* Performance status 0-2
* Left Ventricular Ejection Fraction (LVEF) ≥ 45% within the past 90 days
* diffusing capacity of lung for carbon monoxide (DLCO) ≥ 50%

Exclusion Criteria:

* No overt multiple myeloma, as defined by any of the following:

  * Greater than 30% bone marrow plasmacytosis
  * Extensive (i.e., > 2) lytic lesions
  * Hypercalcemia
* No myocardial infarction, congestive heart failure, or arrhythmia refractory to therapy within the past 6 months
* No prior malignancy except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, adequately treated stage I or II cancer from which the patient is currently in complete response, or any other cancer from which the patient has been disease-free for the past 5 years
* No HIV positivity

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2006-10; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishali Sanchorawala, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston University Cancer Research Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled from the Boston Medical Center Stem Cell Transplant Program between 2006 and 2009.
Pre-assignment Details: A patient enrolled on this study but was withdrawn due to insufficient stem cell yield. His clinical situation changed 5 months later and the investigators believed he would have a better yield so he was enrolled for a second time. Therefore, there were 5 enrollments, but 4 patients.
Groups:
- SCT With Melphalan Conditioning: Mobilization with Filgrastim Stem Cell collection (SCC) Melphalan Conditioning Stem Cell infusion
  filgrastim: 16 mcg/kg daily beginning 3 days prior to SCC through day before final SCC
  melphalan: 70-100 mg/m2/day will be administered intravenously on Days -3 and -2
  Stem Cell Infusion: infusion of previously collected stem cells on Day 0
Period: Overall Study
Arm/Group | SCT With Melphalan Conditioning
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- SCT With Melphalan Conditioning: Mobilization with Filgrastim Stem Cell collection Melphalan Conditioning Stem Cell infusion
  filgrastim: 16 mcg/kg daily beginning 3 days prior to SCC through day before final SCC
  melphalan: 70-100 mg/m2/day will be administered intravenously on Days -3 and -2
  Stem Cell Infusion: infusion of previously collected stem cells on Day 0
Arm/Group | SCT With Melphalan Conditioning
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response Rate
Time Frame: one year
Population: No data were collected or analyzed due to study termination
Arm/Group | SCT With Melphalan Conditioning
Number analyzed (Participants) | 0

2. Secondary Outcome: Predictability of Early Free Light-chain Response for Heme Response
Time Frame: One month
Population: No data were collected or analyzed due to study termination
Arm/Group | SCT With Melphalan Conditioning
Number analyzed (Participants) | 0

3. Secondary Outcome: Organ or Clinical Response
Time Frame: One year
Population: No data were collected or analyzed due to study termination
Arm/Group | SCT With Melphalan Conditioning
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival
Time Frame: life
Population: No data were collected or analyzed due to study termination
Arm/Group | SCT With Melphalan Conditioning
Number analyzed (Participants) | 0

5. Secondary Outcome: Tolerability
Time Frame: 100 days
Population: No data were collected or analyzed due to study termination
Arm/Group | SCT With Melphalan Conditioning
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 100 days
Arm/Group | SCT With Melphalan Conditioning
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCT With Melphalan Conditioning (N=4)
drug reaction (Immune system disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
Toxic Epidermal Necrosis (TEN) (Skin and subcutaneous tissue disorders) | 1 (1)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — related to fluid overload
joint pain (General disorders) | 1 (1) — gout
mucositis (Gastrointestinal disorders) | 2 (2)
voice changes (Gastrointestinal disorders) | 1 (1)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
hypoalbuminemia (Hepatobiliary disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1)
renal insufficiency (Renal and urinary disorders) | 1 (1)
increased creatinine (Renal and urinary disorders) | 1 (1)
hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
febrile neutropenia (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCT With Melphalan Conditioning (N=4)
fatigue (General disorders) | 2 (2)
insomnia (General disorders) | 3 (3)
rigors (General disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (4)
vomiting (Gastrointestinal disorders) | 2 (2)
diarrhea (Gastrointestinal disorders) | 2 (2)
Dehydration (General disorders) | 1 (1)
anorexia (Gastrointestinal disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
sinus tacchycardia (Cardiac disorders) | 2 (2)
peripheral edema (Blood and lymphatic system disorders) | 2 (2)
muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
dizziness (Nervous system disorders) | 1 (1)
seizure (Nervous system disorders) | 1 (1) — grand mal
joint pain (Musculoskeletal and connective tissue disorders) | 2 (2)
bilateral pleural effusions (Respiratory, thoracic and mediastinal disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 1 (1)
elevated ALT (Hepatobiliary disorders) | 1 (1)
hypoalbuminemia (Hepatobiliary disorders) | 3 (3)
elevated alk phos (Hepatobiliary disorders) | 1 (1)
line bleed (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes